CLINICAL TRIAL: NCT03036189
Title: Improving Chronic Illness Management With the Apsaalooke Nation: The Baa Nnilah Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); University of Nevada, Las Vegas (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Suzanne Held, Professor, Montana State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MontanaSU; U01MD010619 (NIH)
Record Dates: First submitted 2017-01-24; First posted 2017-01-30 (Estimated); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: delayed control group design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): There are no devices or drugs used in this trial. The treatment is the same for the intervention arm and the wait-list control arm. The treatment is group trial of 7 meetings designed to improve chronic illness self-management. The name of the treatment is baa nnilah.
  Interventions: Behavioral: baa nnilah
- Wait-list control arm (Experimental): There are no devices or drugs used in this trial. The treatment is the same for the intervention arm and the wait-list control arm. The treatment is group trial of 7 meetings designed to improve chronic illness self-management. The name of the treatment is baa nnilah.
  Interventions: Behavioral: baa nnilah

INTERVENTIONS:
Behavioral: baa nnilah — 7 meetings in the community led by a trained community facilitator

SUMMARY:
This is a group randomized trial of an intervention to improve chronic illness self-management.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 25 years
* AI
* diagnosed with diabetes
* hypertension
* osteoporosis
* liver disease
* chronic lung disease (asthma, chronic bronchitis or emphysema)
* heart disease (coronary artery disease or congestive heart failure)
* stroke (completed cerebrovascular accident with neurologic handicap and normal mentation)
* chronic arthritis

Exclusion Criteria:

* major medical illness that precludes their attendance at 7 meetings
* <25 years of age

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2020-01-29 (Actual); Study Completion 2020-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Held, PhD, Principal Investigator — Montana State University
Locations (1):
- Messengers for Health, Crow Agency, Montana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farivar SS, Cunningham WE, Hays RD. Correlated physical and mental health summary scores for the SF-36 and SF-12 Health Survey, V.I. Health Qual Life Outcomes. 2007 Sep 7;5:54. doi: 10.1186/1477-7525-5-54. PMID 17825096
- [Derived] Hallett J, Feng D, McCormick AKHG, Allen S, Inouye J, Schure M, Holder S, Medicine LO, Held S. Improving Chronic Illness Self-Management with the Apsaalooke Nation: The Baa nnilah Project, a cluster randomized trial protocol. Contemp Clin Trials. 2022 Aug;119:106835. doi: 10.1016/j.cct.2022.106835. Epub 2022 Jun 18. PMID 35724843
- [Derived] Allen S, Held S, Milne-Price S, McCormick A, Feng D, Inouye J, Schure M, Castille D, Howe RB, Pitts M, Keene S, Belone L, Wallerstein N. Community sharing: Contextualizing Western research notions of contamination within an Indigenous research paradigm. Am J Community Psychol. 2022 Mar;69(1-2):145-156. doi: 10.1002/ajcp.12552. Epub 2021 Sep 17. PMID 34534371
- [Derived] Rink E, Knight K, Ellis C, McCormick A, FireMoon P, Held S, Webber E, Adams A. Using Community-Based Participatory Research to Design, Conduct, and Evaluate Randomized Controlled Trials with American Indian Communities. Prev Chronic Dis. 2020 Nov 12;17:E143. doi: 10.5888/pcd17.200099. PMID 33180688

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm | Wait-list Control Arm
Started | 104 | 107
Completed | 69 | 74
Not Completed | 35 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Wait-list Control Arm | Total
Number analyzed (Participants) | 104 | 107 | 211
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: missing data
  years
    number analyzed (Participants) | 101 | 104 | 205
    (all) | 51.71 (13.47) | 52.46 (14.36) | 52.09 (13.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 83 | 152
  Male | 35 | 24 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 104 | 107 | 211
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: SF-12 - Physical Health
Description: The SF-12 is a set of 12 questions regarding function in physical and mental health domains. We changed question 2 to encapsulate moderate activities more applicable to our study population. Activities deleted were bowling and playing golf and activities added were carrying a small child, walking for exercise, or round dancing/push dancing (Native American traditional dances). Participants responded to questions about their physical and mental health, especially regarding the degree of limitation experienced, using varying response categories (i.e., 3, 5, or 6-point Likert scale, or yes/no format). A Physical Component Summary (PCS) score and a Mental Component Summary (MCS) score were computed and normalized based on an algorithm developed by Farivar, Cunningham, and Hays (2007), which used an oblique factor solution for item weights. PCS and MCS scores range from 0 to 100, with higher scores indicating better physical and mental health functioning, respectively.
Time Frame: Intervention group: baseline (T1), up to 1 month (T2), up to 8 months (T3), up to 13 months (T4). WLC group pre-baseline (T1), baseline (T2), up to 1 month (T3), up to 9 months (T4), up to 13 months (T5)
Population: The number of valid data points varied across individuals, as well as by time and by variable within each individual, because participants could 1) miss a data collection but complete subsequent data collection(s) and/or 2) choose not to complete a physical test or a survey question.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm | Wait-list Control Arm
Number analyzed (Participants) | 93 | 94
score on a scale
  T1 | 43.85 (11.18) | 43.64 (9.97)
  T2: number analyzed (Participants) | 74 | 80
  T2 | 45.65 (10.86) | 45.18 (9.42)
  T3: number analyzed (Participants) | 65 | 65
  T3 | 45.56 (11.04) | 44.50 (10.03)
  T4: number analyzed (Participants) | 59 | 67
  T4 | 45.33 (10.53) | 45.26 (9.63)
  T5: number analyzed (Participants) | 0 | 70
  T5 |  | 47.13 (9.51)
Statistical Analysis 1: Comparison: Intervention Arm vs Wait-list Control Arm; Test type: Superiority; p = 0.50, Mixed Models Analysis; Slope = -0.15

2. Primary Outcome: SF-12 - Mental Health
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm | Wait-list Control Arm
Number analyzed (Participants) | 93 | 94
units on a scale
  T1 | 43.85 (11.18) | 43.64 (9.97)
  T2: number analyzed (Participants) | 74 | 80
  T2 | 45.65 (10.86) | 45.18 (9.44)
  T3: number analyzed (Participants) | 65 | 65
  T3 | 45.56 (11.04) | 44.50 (10.03)
  T4: number analyzed (Participants) | 59 | 67
  T4 | 45.33 (10.52) | 45.26 (9.63)
  T5: number analyzed (Participants) | 0 | 70
  T5 |  | 49.30 (10.10)
Statistical Analysis 1: Comparison: Intervention Arm vs Wait-list Control Arm; Test type: Superiority; p = 0.71, Mixed Models Analysis; Slope = .42

3. Secondary Outcome: Patient Health Questionnaire-9
Description: The PHQ-9 is a widely used instrument to measure symptoms of depression. This set of 9 questions asked participants to respond to statements pertaining to their mental health in the preceding 2 weeks. The score range for the instrument is 0-27, with higher scores correlating with higher levels of symptoms of depression. Additionally, there is 1 question, not scored, rating difficulty of problems.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm | Wait-list Control Arm
Number analyzed (Participants) | 103 | 107
units on a scale
  T1 | 5.29 (5.88) | 7.22 (7.47)
  T2: number analyzed (Participants) | 82 | 90
  T2 | 5.43 (6.03) | 6.24 (6.20)
  T3: number analyzed (Participants) | 71 | 75
  T3 | 4.30 (4.87) | 5.50 (5.98)
  T4: number analyzed (Participants) | 69 | 73
  T4 | 5.38 (6.06) | 4.92 (5.70)
  T5: number analyzed (Participants) | 0 | 74
  T5 |  | 4.45 (5.45)
Statistical Analysis 1: Comparison: Intervention Arm vs Wait-list Control Arm; Test type: Superiority; p = 0.83, Mixed Models Analysis; Slope = .12

4. Secondary Outcome: PROMIS Satisfaction With Social Roles and Activities
Description: Patient Reported Outcome Measurement Information System (PROMIS) measure. This 8-item form was used to assess the participant's satisfaction with and ability to participant in social roles and activities, using a 5-point Likert scale. NIH PROMIS measures use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. On the T-score metric a score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population. Higher scores equal more of the concept being measured.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm | Wait-list Control Arm
Number analyzed (Participants) | 102 | 106
units on a scale
  T1 | 53.62 (10.11) | 54.03 (9.62)
  T2: number analyzed (Participants) | 82 | 90
  T2 | 53.26 (10.76) | 53.65 (9.64)
  T3: number analyzed (Participants) | 71 | 75
  T3 | 53.61 (10.01) | 54.05 (9.27)
  T4: number analyzed (Participants) | 69 | 73
  T4 | 53.00 (9.89) | 55.10 (9.36)
  T5: number analyzed (Participants) | 0 | 74
  T5 |  | 55.00 (9.17)
Statistical Analysis 1: Comparison: Intervention Arm vs Wait-list Control Arm; Test type: Superiority; p = 0.58, Mixed Models Analysis; Slope = 0.37

5. Secondary Outcome: PROMIS Self-Efficacy for Managing Symptoms
Description: Patient Reported Outcome Measurement Information System (PROMIS) measure. This 8 item form was used to assess the participant's confidence in their ability to manage symptoms of chronic illness and prevent them from interfering from activities of daily living, using a 5-point Likert scale. NIH PROMIS measures use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. On the T-score metric a score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population. Higher scores equal more of the concept being measured.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm | Wait-list Control Arm
Number analyzed (Participants) | 103 | 106
units on a scale
  T1 | 49.33 (9.64) | 48.15 (9.37)
  T2: number analyzed (Participants) | 82 | 90
  T2 | 48.48 (9.36) | 47.12 (8.34)
  T3: number analyzed (Participants) | 71 | 75
  T3 | 50.45 (8.96) | 48.93 (9.67)
  T4: number analyzed (Participants) | 69 | 73
  T4 | 49.55 (9.86) | 50.61 (9.90)
  T5: number analyzed (Participants) | 0 | 71
  T5 |  | 50.63 (9.94)
Statistical Analysis 1: Comparison: Intervention Arm vs Wait-list Control Arm; Test type: Superiority; p = 0.69, Mixed Models Analysis; Slope = -0.40

6. Secondary Outcome: PROMIS Emotional Support
Description: Patient Reported Outcome Measurement Information System (PROMIS) measure. This 8-item form was used to assess the participant's perception of availability of trusted individuals in their life to provide emotional support, using a 5-point Likert scale. NIH PROMIS measures use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. On the T-score metric a score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population. Higher scores equal more of the concept being measured.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm | Wait-list Control Arm
Number analyzed (Participants) | 103 | 107
units on a scale
  T1 | 52.71 (9.65) | 51.65 (11.09)
  T2: number analyzed (Participants) | 82 | 90
  T2 | 53.31 (8.90) | 53.36 (9.28)
  T3: number analyzed (Participants) | 71 | 75
  T3 | 53.29 (9.09) | 52.32 (10.03)
  T4: number analyzed (Participants) | 69 | 73
  T4 | 53.16 (8.62) | 54.96 (8.35)
  T5: number analyzed (Participants) | 0 | 74
  T5 |  | 53.35 (9.05)
Statistical Analysis 1: Comparison: Intervention Arm vs Wait-list Control Arm; Test type: Superiority; p = 0.60, Mixed Models Analysis; Slope = 0.49

7. Secondary Outcome: PROMIS Positive Affect and Well-being
Description: Patient Reported Outcome Measurement Information System (PROMIS) measure. This 8-item form was used to assess the participant's recent sense of well-being and agreement with positive outlook and experience of life, using a 5-point Likert scale. NIH PROMIS measures use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. On the T-score metric a score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population. Higher scores equal more of the concept being measured.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm | Wait-list Control Arm
Number analyzed (Participants) | 102 | 106
units on a scale
  T1 | 56.32 (7.92) | 56.37 (8.98)
  T2: number analyzed (Participants) | 81 | 90
  T2 | 57.84 (8.18) | 57.37 (8.42)
  T3: number analyzed (Participants) | 71 | 75
  T3 | 57.64 (7.65) | 57.15 (8.37)
  T4: number analyzed (Participants) | 69 | 73
  T4 | 58.50 (8.34) | 58.64 (7.54)
  T5: number analyzed (Participants) | 0 | 59
  T5 |  | 58.35 (6.93)
Statistical Analysis 1: Comparison: Intervention Arm vs Wait-list Control Arm; Test type: Superiority; p = 0.97, Mixed Models Analysis; Slope = -0.03

8. Secondary Outcome: PROMIS Physical Function
Description: Patient Reported Outcome Measurement Information System (PROMIS) measure. This 8 item form was used to assess the function of upper/lower extremities, core, and ability to perform activities of daily living, using a 5-point Likert scale. NIH PROMIS measures use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. On the T-score metric a score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population. Higher scores equal more of the concept being measured.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm | Wait-list Control Arm
Number analyzed (Participants) | 103 | 107
units on a scale
  T1 | 44.94 (8.81) | 45.49 (8.74)
  T2: number analyzed (Participants) | 82 | 90
  T2 | 45.83 (9.08) | 45.55 (8.52)
  T3: number analyzed (Participants) | 71 | 75
  T3 | 45.00 (10.17) | 45.23 (9.28)
  T4: number analyzed (Participants) | 69 | 73
  T4 | 45.91 (10.48) | 44.81 (9.86)
  T5: number analyzed (Participants) | 0 | 74
  T5 |  | 45.82 (8.88)
Statistical Analysis 1: Comparison: Intervention Arm vs Wait-list Control Arm; Test type: Superiority; p = 0.49, Mixed Models Analysis; Slope = 0.45

9. Secondary Outcome: PROMIS Self-efficacy for Managing Emotions
Description: Patient Reported Outcome Measurement Information System (PROMIS) measure. This 8 item form was used to assess the participant's current confidence to manage emotional distress and stressful situations core, using a 5-point Likert scale. NIH PROMIS measures use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. On the T-score metric a score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population. Higher scores equal more of the concept being measured.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm | Wait-list Control Arm
Number analyzed (Participants) | 103 | 107
units on a scale
  T1 | 48.18 (9.13) | 48.28 (9.84)
  T2: number analyzed (Participants) | 82 | 90
  T2 | 50.00 (9.30) | 49.18 (9.93)
  T3: number analyzed (Participants) | 71 | 75
  T3 | 50.15 (8.78) | 49.90 (8.77)
  T4: number analyzed (Participants) | 69 | 73
  T4 | 51.85 (9.37) | 51.70 (8.79)
  T5: number analyzed (Participants) | 0 | 74
  T5 |  | 51.01 (8.45)
Statistical Analysis 1: Comparison: Intervention Arm vs Wait-list Control Arm; Test type: Superiority; p = 0.77, Mixed Models Analysis; Slope = 0.25

10. Secondary Outcome: PROMIS Self-efficacy for Managing Social Interactions
Description: Patient Reported Outcome Measurement Information System (PROMIS) measure. This 4 item form was used to assess the participant's current confidence in being able to access support in processing emotions and health problems, and obtain assistance with transportation and problem solving, using a 5-point Likert scale. NIH PROMIS measures use a T-score metric in which 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. On the T-score metric a score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population. Higher scores equal more of the concept being measured.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm | Wait-list Control Arm
Number analyzed (Participants) | 103 | 106
units on a scale
  T1 | 46.57 (8.57) | 47.44 (9.74)
  T2: number analyzed (Participants) | 82 | 89
  T2 | 47.13 (8.54) | 47.86 (8.99)
  T3: number analyzed (Participants) | 71 | 75
  T3 | 48.57 (9.10) | 47.18 (9.74)
  T4: number analyzed (Participants) | 69 | 73
  T4 | 47.29 (8.94) | 49.20 (8.58)
  T5: number analyzed (Participants) | 0 | 71
  T5 |  | 49.17 (8.60)
Statistical Analysis 1: Comparison: Intervention Arm vs Wait-list Control Arm; Test type: Superiority; p < .05, Mixed Models Analysis; Slope = 0.54

11. Secondary Outcome: Patient Activation Measure
Description: PAM assesses self-management related health knowledge, skills, and confidence. Developed by Insignia Health as a 22-item measure and shortened to 13 questions, with the short form validated to assess patient knowledge, skill and confidence for self-management of health conditions. We used the 13-item measure. Insignia Health's proprietary survey scoring algorithm produces a PAM Score along an empirical, interval-level scale from 0-100 with higher scores indicating higher patient activation.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention Arm | Wait-list Control Arm
Number analyzed (Participants) | 104 | 107
units on a scale
  T1 | 69.31 (17.73) | 65.50 (16.41)
  T2: number analyzed (Participants) | 82 | 90
  T2 | 67.53 (21.22) | 70.61 (19.66)
  T3: number analyzed (Participants) | 71 | 75
  T3 | 68.47 (20.88) | 71.67 (17.97)
  T4: number analyzed (Participants) | 66 | 73
  T4 | 67.05 (17.91) | 71.57 (18.59)
  T5: number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Intervention Arm vs Wait-list Control Arm; Test type: Superiority; p = 0.40, Mixed Models Analysis; Slope = 1.99

12. Secondary Outcome: Modified Timed Up and Go
Description: The TUG test is physical test that assists in screening and measurement of balance deficits in older adults, which correlates with increased fall risk, and has been validated across populations. In this physical test, participants sit in a chair with feet flat on the ground and back against the chair. A timer is started as they leave the chair, and continues as they pace 3 meters, execute a 180 degree turn and just as they touch the chair again, the timer is stopped. Due to an error in communication between a consultant who assisted with this measure and the research team, the distance that individuals walked during this test was modified from 3 m to 10 m, therefore prior validation data may not apply.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intervention Arm | Wait-list Control Arm
Number analyzed (Participants) | 99 | 105
seconds
  T1 | 20.83 (5.43) | 20.39 (5.30)
  T2: number analyzed (Participants) | 74 | 80
  T2 | 19.26 (5.08) | 19.34 (4.31)
  T3: number analyzed (Participants) | 63 | 67
  T3 | 17.18 (5.51) | 18.70 (7.30)
  T4: number analyzed (Participants) | 45 | 41
  T4 | 18.42 (4.27) | 18.26 (3.79)
  T5: number analyzed (Participants) | 0 | 53
  T5 |  | 19.06 (4.58)
Statistical Analysis 1: Comparison: Intervention Arm vs Wait-list Control Arm; Test type: Superiority; p = 0.07, Mixed Models Analysis; Slope = 1.05

13. Secondary Outcome: Modified Balance Error Scoring System
Description: The original Balance Error Scoring System (BESS) involved firm and padded surface balance testing in 3 positions, to assess static balance and was validated across study populations. The mBESS only utilizes firm surface data and demonstrated better intertester reliability and validity. During this physical test, a staff member counts how many times participants help themselves to regain balance in 20 seconds. The mBESS involved 3 positions, depicted below. Participants stood with hands on hips and eyes closed, balancing for 20 s in 3 standing positions: a double-leg stance, a single-leg stance, and tandem stance. Test observers counted up to 10 errors per stance, including opening eyes, taking hands off hips, stepping, putting a hand out to a chair or wall, or making other large corrections, which led to a stance score ranging from 0 to 10 with a maximum total of 30. Participants who could not complete a position for balance reasons, were given a score of 10.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: total number of errors over three trials
Arm/Group | Intervention Arm | Wait-list Control Arm
Number analyzed (Participants) | 90 | 106
total number of errors over three trials
  T1 | 13.41 (6.33) | 13.81 (6.60)
  T2: number analyzed (Participants) | 78 | 84
  T2 | 14.17 (7.22) | 12.68 (6.59)
  T3: number analyzed (Participants) | 60 | 68
  T3 | 15.30 (10.26) | 11.91 (10.57)
  T4: number analyzed (Participants) | 70 | 74
  T4 | 20.96 (8.87) | 21.03 (9.44)
  T5: number analyzed (Participants) | 0 | 53
  T5 |  | 13.38 (6.94)
Statistical Analysis 1: Comparison: Intervention Arm vs Wait-list Control Arm; Test type: Superiority; p = 0.84, Mixed Models Analysis; Slope = 2.00

14. Secondary Outcome: 6-minute Walk
Description: Serves as a corollary for physical function and cardiovascular performance.Participants walked at a comfortable pace for six minutes and their distance was recorded in feet.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Intervention Arm | Wait-list Control Arm
Number analyzed (Participants) | 97 | 98
feet
  T1 | 1260.23 (287.70) | 1298.85 (265.40)
  T2: number analyzed (Participants) | 68 | 76
  T2 | 1336.75 (273.48) | 1358.96 (323.35)
  T3: number analyzed (Participants) | 56 | 57
  T3 | 1060.11 (603.53) | 1283.54 (449.10)
  T4: number analyzed (Participants) | 43 | 43
  T4 | 1312.84 (379.76) | 1334.98 (284.74)
  T5: number analyzed (Participants) | 0 | 53
  T5 |  | 1287.08 (320.25)
Statistical Analysis 1: Comparison: Intervention Arm vs Wait-list Control Arm; Test type: Superiority; p = 0.64, Mixed Models Analysis; Slope = -23.01

ADVERSE EVENTS:
Time Frame: through study completion, which was 2 years and 4 months long
Arm/Group | Intervention Arm | Wait-list Control Arm
All-Cause Mortality (participants affected / at risk) | 5/104 | 1/107
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/107
Other Adverse Events (participants affected / at risk) | 0/104 | 0/107

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/89/NCT03036189/Prot_001.pdf
  • Statistical Analysis Plan (2022-08-23): https://cdn.clinicaltrials.gov/large-docs/89/NCT03036189/SAP_002.pdf
  • Informed Consent Form (2017-08-20): https://cdn.clinicaltrials.gov/large-docs/89/NCT03036189/ICF_000.pdf